CLINICAL TRIAL: NCT03600857
Title: Medical Termination of Pregnancy From Day 85 to Day 153 of Gestation: A Randomized Comparison Between Administration of the Initial Dose of Misoprostol at Home or in the Clinic
Brief Title: Medical Termination of II Trimester Pregnancy
Acronym: PRIMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kristina Gemzell Danielsson, Professor, Överläkare, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: WP2018
Record Dates: First submitted 2018-06-02; First posted 2018-07-26 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Unwanted Pregnancy
Keywords: medical abortion; mifepristone; misoprostol; home use

STUDY DESIGN:
Intervention Model Description: Open label, multicentre, RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home administration (Experimental): Home administration of 0.8 mg misoprostol pv
  Interventions: Other: Home administration of misoprostol
- Hospital administration (No Intervention): Hospital administration of 0.8 mg misoprostol pv

INTERVENTIONS:
Other: Home administration of misoprostol — First dose of misoprostol administration at home
  Arms: Home administration

SUMMARY:
The objective of this study is to compare two groups of women requiring termination of pregnancy from the gestational age of 85 days. All women will receive Mifepristone during their first visit to the out-patient ward. One group of women will receive Misoprostol to administer the first dose (vaginally) at home and 2 hours later they will be admitted to the in-patient ward. They will be informed to present earlier if they start bleeding or experience pain corresponding to more than normal menstrual cramping.

The other group will receive the first dose of Misoprostol (vaginally) when admitted in the in-patient ward (usually in the morning) according to current practice.

ELIGIBILITY:
Inclusion Criteria:

* Women aged >/= 18 years requesting a termination of pregnancy, for social, medical or foetal indications
* gestational age 85 - 153 days (with ultrasonography),
* willing and able to understand and participate after the study has been explained, with good understanding of Swedish or English language,
* general good health,
* single intra-uterine pregnancy,

Exclusion Criteria:

* do not wish to participate or unable to communicate in Swedish or English.
* non-viable pregnancy (confirmed by ultrasonography).
* a history or evidence of disorders that represent a contraindication to the use of Mifepristone or Misoprostol (adrenal pathology, steroid dependent cancer, porphyria, known allergy to the medication).
* any pre-existing health conditions for whom the execution of a medical abortion as judged by the investigator could compromise their condition (Examples of health conditions of concern are: severe anaemia, severe asthma, haemorrhagic disorders, treatment with anticoagulants or corticoids, severe cardiac disease or hypertension, severe liver disease, severe kidney disease or severe psychiatric disorders).
* Fetal malformation that may impact time-to-expulsion (such as hydrocephalus, hydrops/edema) or a duplex pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of women treated as day care patients | 9 hours from admission to the out patient clinic
  No overnight hospitalization required.

SECONDARY OUTCOMES:
induction-to-abortion interval | From first dose of misoprostol until the expulsion of the foetus or surgical intervention whichever comes first assessed up to 7 days of induction
  time in minutes
Time spent in hospital | From admission until discharge up to 2 weeks FU
  Duration of time in hospital in hours
the success rate of the termination of pregnancy at 24 hours | At 24 hours from first dose of misoprostol
  success will be defined as the expulsion of the foetus
Dose of misoprostol | From the first dose to the last dose until 2 weeks FU
  Total dose
Administration of misoprostol | From the first dose to the last dose until 2 weeks FU
  Number of doses
Surgical intervention | From the administration of mifepristone until 2 weeks FU
  surgical interventions for incomplete or retained placenta (evacuation rates)
ncidence of Treatment-Emergent Adverse Events [Safety and Tolerability | From the administration of mifepristone until 2 weeks FU
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0visit
Acceptability | At follow up two weeks after abortion
  Acceptability with allocated treatment (evaluated by two pretested questions)
Painscores | From the administration of mifepristone until 2 weeks FU
  maximal pain score during the abortion measured on a 10mm visual analogue scale from 1 to 10mm

OTHER OUTCOMES:
Premature admissions | Time form Intake of mifepristone until 54 hours
  number of women who need to be admitted to the hospital earlier prior to planned admission and for which reasons will be registered.

CONTACTS AND LOCATIONS:
Locations (4):
- Sweden (4):
  - The Department of Obstetrics and Gynaecology at Danderyd Hospital:, Stockholm, Danderyd
  - WHOcentre, Karolinska University Hospital, Stockholm, Solna
  - Clinics of Obstetrics and Gynaecology at: The Department of Gynecology and reproductive Medicine at Östra sjukhuset, Sahlgrenska University Hospital,, Gothenburg
  - The Department of Obstetrics/Gynaecology, Stockholm South General Hospital (Södersjukhuset),, Stockholm

IPD SHARING:
Plan to Share IPD: No